CLINICAL TRIAL: NCT03224325
Title: A Randomized, Investigator and Subject Blinded, Sponsor Unblinded Placebo-Controlled Phase I Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Escalating Multiple Doses of TAK-831 in Healthy Subjects
Brief Title: A Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Escalating Multiple Doses of TAK-831 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-831-1005
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Results first posted 2019-11-19 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo (Pooled) (Other): TAK-831 placebo-matching suspension, orally, once daily (QD) for up to Day 16.
  Interventions: Drug: Placebo
- TAK-831 100 mg (Experimental): TAK-831 100 mg, tablets, orally, QD on Days 1 and 3 to 16.
  Interventions: Drug: TAK-831 Tablet T2
- TAK-831 300 mg (Experimental): TAK-831 300 mg, tablets, orally, QD on Days 1 and 3 to 16.
  Interventions: Drug: TAK-831 Tablet T2
- TAK-831 600 mg (Experimental): TAK-831 600 mg, tablets, orally, QD on Days 1 and 3 to 16.
  Interventions: Drug: TAK-831 Tablet T2
- TAK-831 15 mg (Experimental): TAK-831 15 mg, suspension, orally, multiple doses (MD) daily, on Days 1 and 3 to 16.
  Interventions: Drug: TAK-831 Suspension
- TAK-831 800 mg (Experimental): TAK-831 800 mg, suspension, orally, QD on Day 1, MD on Days 3 to 16.
  Interventions: Drug: TAK-831 Suspension
- TAK-831 1200 mg (Experimental): TAK-831 1200 mg, suspension, orally, QD on Day 1, MD on Days 3 to 16.
  Interventions: Drug: TAK-831 Suspension

INTERVENTIONS:
Drug: TAK-831 Tablet T2 — Tak-831 tablets.
  Arms: TAK-831 100 mg; TAK-831 300 mg; TAK-831 600 mg
Drug: Placebo — TAK-831 placebo-matching suspension.
  Arms: Placebo (Pooled)
Drug: TAK-831 Suspension — TAK-831 Suspension.
  Arms: TAK-831 1200 mg; TAK-831 15 mg; TAK-831 800 mg

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of TAK-831 when administered as multiple oral doses at escalating dose levels in healthy participants.

DETAILED DESCRIPTION:
This study is a randomized, investigator and participant blinded, sponsor unblinded, placebo-controlled, study of the safety, tolerability and pharmacokinetics of TAK-831 in up to 48 healthy volunteers, with 8 subjects in each of the 6 cohorts.

In each cohort, participants will be randomized in a 3:1 ratio to receive TAK-831 or placebo. Two formulations, oral suspension and tablet will be tested in this study. Both blood and cerebrospinal fluid (CSF) samples will be collected from selected cohorts (CSF cohorts); for the rest of the cohorts, only blood samples will be collected (non-CSF cohorts).

This single-center trial will be conducted in the United States. The overall time to participate in this study is 58 days. Participants will make multiple visits to the clinic, and 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has at least 45 kg weight and has a body mass index (BMI) from 18.0 to 30.0 kilogram per square meter (kg/m^2), inclusive at Screening.
2. The participant is a healthy male or female not of childbearing potential adult who is aged 18 to 55 years, inclusive, at the time of informed consent and first study drug dose.
3. A male participant who is non-sterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 90 days plus half-lives (95 days) after last study drug dose.
4. A female participant with no childbearing potential, defined as a participant that has been surgically sterilized (hysterectomy, bilateral oophorectomy or tubal ligation) or who is postmenopausal (defined as continuous amenorrhea of at least 12 months and follicle stimulating hormone [FSH] greater than [>] 40 international unit per liter [IU/L]).

Exclusion Criteria:

1. Has a positive urine drug result for drugs of abuse (defined as any illicit drug use) at Screening or Check-in.
2. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as >3 drinks per day) within 5 years before the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. (1 drink=12 ounce [oz]. beer=5 oz. wine=1.5 oz. liquor.)
3. Has a QT interval with Fridericia's correction method (QTcF) >450 milliseconds (ms) (male participants) or >470 ms (female participants) or PR outside the range of 120 to 220 ms, confirmed with 1 repeat testing, at the Screening Visit or Check-in. When triplicate electrocardiogram (ECG) assessments are collected, the mean of the 3 QTcF and PR values should be used to assess this criterion.
4. Has a positive test result for hepatitis B surface antigen (HBsAg), anti- human chorionic gonadotropin (HCV), or human immunodeficiency virus (HIV) antibody/antigen at Screening.
5. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days before Check-in. Cotinine test is positive at Screening or Check-in.
6. Has poor peripheral venous access.
7. Has donated or lost 450 milliliter (mL) or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days before the first dose of study medication.
8. Has a Screening or Check-in abnormal (clinically significant) ECG. Entry of any participant with an abnormal (not clinically significant) ECG must be approved and documented by signature by the principal investigator or designee.
9. Has a supine blood pressure outside 90 to 140 millimeter of mercury (mm Hg) for systolic and 50 to 90 mm Hg for diastolic, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in.
10. Has a resting heart rate outside 40 to 100 beats per minute confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (heart rate from the ECG does not apply).
11. Has a risk of suicide according to the Investigator's clinical judgment (example, per Columbia-Suicide Severity Rating Scale [C-SSRS]), or has scored "yes" on item 4 or item 5 of the Suicidal Ideation section of the C-SSRS, if this ideation occurred in the past 6 months, or "yes" on any item of the Suicidal Behavior section, except for the "Non-Suicidal Self-Injurious Behavior", if this behavior occurred in the past 2 years.

    Additional Exclusion Criteria for Cohort(s) with cerebrospinal fluid (CSF) Collection:
12. Has had CSF collection performed within 30 days before Check-in.
13. Has a history of clinically significant back pain and/or injury.
14. Has local infection at the puncture site.
15. Has thrombocytopenia or other suspected bleeding tendencies noted before procedure.
16. Has developed signs and symptoms of spinal radiculopathy, including lower extremity pain and paresthesia.
17. Has any focal neurological deficit that might suggest an increase in intracranial pressure.
18. Has any abnormal findings on ophthalmological assessment/fundoscopy suggestive of raised intracranial pressure (that is, optic disc swelling/edema; (uncontrolled) hypertensive retinopathy).
19. Suffers regularly from moderate to severe headaches requiring analgesics.
20. Has lower spinal malformations (on physical examination or lumbar spine radiography), local spinal infection, or other abnormalities that would exclude lumbar puncture (LP).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2018-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- California Clinical Trials Medical Group/PAREXEL, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 21-Jul-2017 to 9-Sep-2018.
Pre-assignment Details: Healthy volunteers were enrolled in a 1:3 ratio to receive placebo or TAK-831 in 6 cohorts.
Groups:
- Placebo (Pooled): TAK-831 placebo-matching suspension, orally, once daily (QD) on Days 1 and 3 to 16.
Period: Overall Study
Arm/Group | Placebo (Pooled) | TAK-831 100 mg | TAK-831 300 mg | TAK-831 600 mg | TAK-831 15 mg | TAK-831 800 mg | TAK-831 1200 mg
Started | 13 | 6 | 6 | 6 | 6 | 6 | 7
Completed | 12 | 6 | 6 | 5 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo (Pooled): TAK-831 placebo-matching suspension, orally, QD on Days 1 and 3 to 16.
- Total: Total of all reporting groups
Arm/Group | Placebo (Pooled) | TAK-831 100 mg | TAK-831 300 mg | TAK-831 600 mg | TAK-831 15 mg | TAK-831 800 mg | TAK-831 1200 mg | Total
Number analyzed (Participants) | 13 | 6 | 6 | 6 | 6 | 6 | 7 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (10.96) | 35.7 (7.61) | 30.0 (6.99) | 42.8 (7.63) | 45.2 (5.56) | 35.5 (6.63) | 37.0 (9.09) | 38.0 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 6
  Male | 12 | 6 | 6 | 5 | 5 | 4 | 6 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 1 | 2 | 2 | 4 | 16
  Not Hispanic or Latino | 11 | 3 | 4 | 5 | 4 | 4 | 3 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Black or African American | 5 | 3 | 0 | 2 | 0 | 2 | 0 | 12
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  White | 5 | 3 | 5 | 4 | 6 | 3 | 7 | 33
  Multiracial | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 6 | 6 | 6 | 6 | 6 | 7 | 50
Weight [Mean (Standard Deviation); unit: kg] | 81.21 (12.06) | 82.58 (8.443) | 77.40 (10.22) | 84.95 (11.85) | 77.67 (8.823) | 82.07 (13.18) | 75.56 (10.78) | 80.25 (10.81)
Height [Mean (Standard Deviation); unit: cm] | 176.8 (7.87) | 177.3 (7.47) | 176.8 (9.66) | 175.8 (6.85) | 173.3 (10.42) | 173.2 (10.03) | 171.1 (8.30) | 175.1 (8.36)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=Weight/Height^2.
  kg/m^2 | 26.00 (3.028) | 26.50 (1.761) | 24.83 (3.312) | 27.33 (2.338) | 25.67 (2.066) | 27.17 (2.483) | 25.86 (3.388) | 26.16 (2.691)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Treatment-Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an AE with an onset that occurs after receiving study drug.
Time Frame: Baseline up to 30 days after the last dose (Up to 48 days)
Population: Safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Pooled) | TAK-831 100 mg | TAK-831 300 mg | TAK-831 600 mg | TAK-831 15 mg | TAK-831 800 mg | TAK-831 1200 mg
Number analyzed (Participants) | 13 | 6 | 6 | 6 | 6 | 6 | 7
percentage of participants | 69.2 | 83.3 | 100.0 | 66.7 | 100.0 | 100.0 | 42.9

2. Primary Outcome: Percentage of Participants Who Met the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Postdose
Description: Clinical Laboratory parameters included tests for chemistry, hematology and urinalysis. Markedly abnormal values during treatment period were categorized as: alanine aminotransferase (ALT)>3.0 U/L*upper limit of normal(ULN), albumin<25 g/L, alkaline phosphatase >3.0 U/L*ULN, aspartate aminotransferase >3.0 U/L*ULN, bilirubin >3.42 umol/L creatinine >177umol/L, gamma glutamyl transferase (GGT) >3 U/L*ULN, glucose <2.8 mmol/L, >19.4 mmol/L, potassium<3 mmol/L, >6 mmol/L, sodium <130 mmol/L, >150 mmol/L, protein <0.8 g/L,* lower limit of normal (LLN), >1.2 g/L*ULN, erythrocytes <0.8 (10^12/L)*LLN, >1.2 (10^12/L)*ULN, hematocrit (%) <0.8*LLN, >1.2*ULN, hemoglobin <0.8 g/L*LLN, >1.2 g/L*ULN, leukocytes <0.5 (10^9/L)*LLN, >1.5 (10^9/L)*ULN, platelets <75(10^9/L), >600(10^9/L). Only categories with values have been reported.
Time Frame: Baseline up to 30 days after the last dose (Up to 48 days)
Population: Safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Pooled) | TAK-831 100 mg | TAK-831 300 mg | TAK-831 600 mg | TAK-831 15 mg | TAK-831 800 mg | TAK-831 1200 mg
Number analyzed (Participants) | 13 | 6 | 6 | 6 | 6 | 6 | 7
percentage of participants | 0 | 0 | 16.7 | 0 | 16.7 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Met the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Postdose
Description: Vital signs included temperature, pulse rate and blood pressure. Markedly abnormal values during treatment period were categorized as: Pulse Rate (beats/min) <50->120, Systolic Blood Pressure (SBP) (mmHg) <85->180, Diastolic Blood Pressure (DBP) (mmHg) <50->110 and Temperature (degree centigrades) <35.6- >37.7.
Time Frame: Baseline up to 30 days after the last dose (Up to 48 days)
Population: Safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Pooled) | TAK-831 100 mg | TAK-831 300 mg | TAK-831 600 mg | TAK-831 15 mg | TAK-831 800 mg | TAK-831 1200 mg
Number analyzed (Participants) | 13 | 6 | 6 | 6 | 6 | 6 | 7
percentage of participants | 92.3 | 83.3 | 100 | 66.7 | 83.3 | 66.7 | 42.9

4. Primary Outcome: Percentage of Participants Who Met the Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) Parameters at Least Once Postdose
Description: A 12-lead ECG was performed. Markedly abnormal values during treatment period were categorized as: ECG Mean Heart Rate (beats/min) <50->120, PR Interval, Aggregate (msec) <=80->=200, QRS Duration, Aggregate (msec) <=80->=180, QT Interval, Aggregate (msec) <=300->=460, QTcF Interval, Aggregate (msec) <=300->=500 OR >=30 change from baseline and >=450 milliseconds.
Time Frame: Baseline up to 30 days after the last dose (Up to 48 days)
Population: Safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Pooled) | TAK-831 100 mg | TAK-831 300 mg | TAK-831 600 mg | TAK-831 15 mg | TAK-831 800 mg | TAK-831 1200 mg
Number analyzed (Participants) | 13 | 6 | 6 | 6 | 6 | 6 | 7
percentage of participants | 38.5 | 83.3 | 66.7 | 16.7 | 66.7 | 66.7 | 42.9

5. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-831
Time Frame: 0.5 hours pre-dose and at multiple timepoint (Up to 24 hours) post-dose on Day 1
Population: The PK set included all participants from the safety set who had at least 1 measurable post dose TAK-831 plasma concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-831 100 mg | TAK-831 300 mg | TAK-831 600 mg | TAK-831 15 mg | TAK-831 800 mg | TAK-831 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 7
ng/mL | 242.2 (101.98) | 566.7 (233.48) | 1008.8 (387.83) | 140.0 (58.43) | 1721.2 (558.38) | 2682.9 (945.83)

6. Secondary Outcome: Cmax ss: Maximum Observed Steady-state Plasma Concentration During a Dosing Interval for TAK-831
Time Frame: 0.5 hours pre-dose and at multiple timepoint (Up to 24 hours) post-dose on Day 16
Population: The PK set included all participants from the safety set who had at least 1 measurable post dose TAK-831 plasma concentration with data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-831 100 mg | TAK-831 300 mg | TAK-831 600 mg | TAK-831 15 mg | TAK-831 800 mg | TAK-831 1200 mg
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 7
ng/mL | 220.8 (99.52) | 528.2 (125.48) | 1494.0 (325.78) | 165.0 (51.26) | 2048.3 (610.39) | 3351.7 (1125.62)

7. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-831
Time Frame: 0.5 hours pre-dose and at multiple timepoint (Up to 24 hours) post-dose on Days 1 and 16
Population: The PK set included all participants from the safety set who had at least 1 measurable post dose TAK-831 plasma concentration. Number analyzed is the number of participants with data available for analysis for the given timepoint.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | TAK-831 100 mg | TAK-831 300 mg | TAK-831 600 mg | TAK-831 15 mg | TAK-831 800 mg | TAK-831 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 7
hours (hr)
  Day 1 | 0.760 [0.50 to 1.50] | 1.265 [1.02 to 1.63] | 1.775 [1.00 to 4.00] | 0.500 [0.50 to 0.50] | 2.000 [1.92 to 4.03] | 2.020 [0.52 to 2.07]
  Day 16: number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 6
  Day 16 | 0.500 [0.50 to 2.15] | 1.475 [0.98 to 2.00] | 2.000 [1.00 to 2.07] | 0.500 [0.48 to 0.50] | 2.000 [1.00 to 2.00] | 2.000 [1.00 to 2.02]

8. Secondary Outcome: AUC0-24: Area Under the Plasma Concentration-time Curve During a Dosing Interval for TAK-831
Time Frame: 0.5 hours pre-dose and at multiple timepoint (Up to 24 hours) post-dose on Days 1 and 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | TAK-831 100 mg | TAK-831 300 mg | TAK-831 600 mg | TAK-831 15 mg | TAK-831 800 mg | TAK-831 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 7
hr*ng/mL
  Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
  Day 1 | 547.7 (129.20) | 1660.6 (111.26) | 3715.0 (1209.59) | 212.7 (72.43) | 7732.2 (474.07) | 10053.7 (2254.51)
  Day 16 | 558.5 (269.85) | 1987.1 (381.65) | 5078.5 (1085.34) | 273.0 (79.74) | 8985.3 (1616.82) | 11818.3 (3355.60)

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after the last dose (Up to 48 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
  Safety set included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo (Pooled) | TAK-831 100 mg | TAK-831 300 mg | TAK-831 600 mg | TAK-831 15 mg | TAK-831 800 mg | TAK-831 1200 mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 9/13 | 5/6 | 6/6 | 4/6 | 6/6 | 6/6 | 3/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Pooled) (N=13) | TAK-831 100 mg (N=6) | TAK-831 300 mg (N=6) | TAK-831 600 mg (N=6) | TAK-831 15 mg (N=6) | TAK-831 800 mg (N=6) | TAK-831 1200 mg (N=7)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 5 | 4 | 5 | 3 | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 1 | 4 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 0 | 5 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 1
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 3 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Medical device site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI may publish results of the study following the publication of results by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT03224325/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT03224325/SAP_001.pdf